CLINICAL TRIAL: NCT01817361
Title: Oral Health and People With Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hon K. Yuen, PhD, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 1R21DE017360-01A2 (NIH)
Record Dates: First submitted 2013-03-12; First posted 2013-03-25 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Systemic Sclerosis
Keywords: oral health
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The public health impact of this study will be the application of the greater understanding of the oral health status, oral health related behaviors, and quality of life of patients with systemic sclerosis (scleroderma or SSc). It is hoped that risks and protective factors can be identified to be associated with the oral health status of adults with systemic sclerosis,leading to the development of interventions for improved oral health in this population,and providing the basis for a larger study of oral health problems of adults with systemic sclerosis.

DETAILED DESCRIPTION:
The broad, long-term objective of our proposed research is to understand the oral health status, oral health-related behaviors, and quality of life in the US population of patients with systemic sclerosis (scleroderma or SSc). SSc is a rare, progressive connective tissue disease that affects predominately women (3.8:1) with a higher risk of the severe form among African-Americans. SSc adults experience manifestations of the systemic disease that include microstomia, xerostomia, and impaired manual dexterity. The two specific aims of this study are: 1) to characterize the oral health status of adults with SSc, and 2) to determine the SSc disease specific manifestations (microstomia, xerostomia, and manual dexterity impairments) that are associated with the severity of oral health problems and oral health-related quality of life among adults with SSc. This first study of US adults with SSc is a cross-sectional survey of 250 adults with SSc in South Carolina. This population is 25% African-American which is similar to the racial distribution of SSc in the US adult population. Data collection includes information on: oral health status (periodontal, dental, mucosal and microbial), oral manifestations of SSc (size of oral aperture, severity of oral dryness, and manual dexterity for oral hygiene), and oral health-related behaviors and quality of life. The oral health status of the South Carolina SSc population will be compared to that of the adult US population based on an analysis of corresponding measures using the National Health and Nutrition Examination Survey 1999-2002 data. Multivariable regression modeling will be used to evaluate hypothesized risk and protective factors that are associated with oral health status in adults with SSc. Results of this study in South Carolina will be used in regional efforts for the development of interventions for improved oral health status of adults with SSc. Second, these results will provide the basis for a larger US study of oral health problems of adults with SSc.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SSc according to American College of Rheumatology criteria, and participants are 18 years of age or older at the time of invitation to the study.

Exclusion Criteria:

* participants who require antibiotic medication before dental treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with systemic sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Oral Health Status as measured by periodontal disease | baseline to 2.5 years
  Periodontal disease will be measured by the loss of attachment of 4mm or more at one or more sites. The number of subjects presenting with periodontal disease will be reported.
Oral Health Status as measured by untreated dental decay | baseline to 2.5 years
  Measure description: Untreated dental decay will be determined by either the presence of coronal caries quantified by using the D component of the DMFS Index. The DMFS Index quantifies the dental caries experience by the number of decayed (D), missing (M), and filled (F) dental surfaces (S). OR by identification of the presence of root caries, which will be recorded following the Centers for Disease Control and Prevention (CDC), National Health and Nutrition Examination Survey (NHANES) 1999-2002 protocol (https://wwwn.cdc.gov/nchs/data/nhanes3/manuals/dental.pdf). The protocol includes a half-mouth examination is done using a quadrant from each the maxillary and mandibular regions for a maximum of 14 teeth (third molars excluded). For each participant, the quadrant selection is randomly generated by the computer program. The number of subjects presenting with untreated dental decay will be reported
Oral Health Status as measured by number of subjects with missing teeth | baseline to 2.5 years
  Measure description: The number of missing teeth (T) is quantified using the D (decayed) component of the DMFT Index. The DMFT Index quantifies the dental caries experience by the number of decayed (D), missing (M), and filled (F) teeth (T). The number of subjects presenting with missing teeth will be reported.
Oral Health Status as measured by the mean size of the aperture among subjects | baseline to 2.5 years
  Size of oral aperture will be measured by both the maximum incisor and maximum lip aperture to define size of oral aperture. Maximum incisor aperture (i.e., interincisal distance) will be the vertical distance in millimeters from the bottom of the maxillary right central incisor to the top of the mandibular incisor when the participants open their mouth as wide as possible. Maximum lip aperture (i.e., interlabial distance) is the vertical distance in millimeters from the bottom of the top lip to the top of the bottom lip when the participants open their mouth as wide as possible. An average of three successive trials for each oral aperture measurement will be used. Microstomia is defined as the interlabial distance <45 mm or the interincisal distance <40 mm. Further, moderate microstomia is when the interincisal distance is between 31-40 mm, and severe microstomia is when the interincisal distance is less than 30 mm. The mean size of the aperture among subjects will be reported.
Oral Health Status as measured by perceived dryness | baseline to 2.5 years
  The presence or absence of oral dryness will be quantified using the perceived oral dryness index. The subjective experience of dry mouth will be assessed by asking each participant about the amount of saliva in the mouth and about dry mouth during meals. Four self-reported questions developed by Fox et al .have been shown to significantly correlate with unstimulated salivary output and salivary flow rates. A "yes" response to one or more of the following four questions is considered positive for xerostomia: (1) Does your mouth feel dry when eating a meal? (2) Do you sip liquids to aid in swallowing dry foods? (3) Do you have difficulties swallowing any foods? (4) Does the amount of saliva in your mouth seem to be too little? The number of subjects presenting with perceived dryness will be reported.
Oral Health Status as measured by residual saliva level | baseline to 2.5 years
  The severity of oral dryness is quantified by measuring the residual saliva levels at the lower inner lip. The lower inner lip location for residual saliva is suggested as a sensitive measure of oral dryness. Participants are instructed not to eat or drink for at least one hour before the measurement. The residual saliva in this location will be collected using a standard SialopaperTM strip (Ora Flow Inc) which is held with a cotton plier. Participants are instructed to dry swallow and the mucosal surface of their lower inner lip as indicated by DiSabato-Mordarski & Kleinberg will be immediately touched with the SialopaperTM strip in a dipstick fashion for 5 seconds. The amount of absorbed saliva (in μl) on the strip will be measured electronically with the Periotron 8000® micro-moisture meter (Ora Flow Inc). The score will range from 0-200. The mean residual saliva level among subjects will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Hon K Yuen, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States